CLINICAL TRIAL: NCT02008708
Title: Microfinance Intervention to Improve Health of Trauma Survivors in DRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Nancy Glass, Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01MD006075 (NIH); R01MD006075 (NIH)
Record Dates: First submitted 2013-10-07; First posted 2013-12-11 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Mental Disorders; Multiple Trauma
Keywords: Health; Microfinance
MeSH Terms: conditions — Mental Disorders; Multiple Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Livestock microfinance (Experimental): Participants randomized to the microfinance intervention receive a female pig loan with ongoing support to manage health and care of the pig by trained agents.
  Interventions: Behavioral: Livestock Microfinance
- Delayed Control Group (Active Comparator): Participants randomized to delayed control group receives pig loan 12 months after the intervention group
  Interventions: Other: Delayed Control Group

INTERVENTIONS:
Behavioral: Livestock Microfinance — Participants randomized to the microfinance group receive the pig loan.
  Arms: Livestock microfinance
Other: Delayed Control Group — Participants enrolled in delayed control receive their pig loan 12 months after the intervention group.
  Arms: Delayed Control Group

SUMMARY:
The objective is to test the effectiveness of a village-led microfinance program, Pigs for Peace, on health, household economic stability, and reintegration of trauma survivors to family and community.

The five-year experimental trial will use mixed-methods to address the following aims:

1. Determine the effectiveness of a village-led microfinance program on participants health and reintegration in intervention households compared to participants in delayed control households. Health and reintegration will be measured at baseline and six, twelve, and 18-months post-baseline using self-report in both intervention and delayed control groups. We hypothesize that at six, twelve and 18 months post-baseline participants in intervention households will have improved health and increased reintegration to families in comparison to participants in control households.
2. Determine the effectiveness of a village-led microfinance program on household economic stability in intervention households compared to delayed control villages. Household economic stability will be measured at baseline and six, twelve and 18 months post- baseline using self-report in both intervention and control households. We hypothesize that at six, twelve and 18-months post-baseline the intervention households will have improved household economic stability in comparison to control households.
3. Examine the role of a village-led microfinance program on village-level health, economics, stigma and reintegration of survivors and their families in intervention and delayed control villages. Village members (n=5 in each village, n=50 total) will complete a baseline and 18 month post-baseline qualitative interview to examine the role of microfinance on village-level health, economics, stigma and reintegration in both intervention and control households.

DETAILED DESCRIPTION:
Mobutu Sese Seko's government of "Kleptocracy" collapsed in 1997 after 30 years of oppression. The new nation that emerged, the Democratic Republic of Congo (DRC), remains an all-to-potent reminder of how human rights violations, and their related health and economic impacts, can devastate individuals, families and communities. The genocide in neighboring Rwanda, coupled with the collapse of the Mobutu government, has spawned two wars and over a decade of warfare throughout the region, resulting in millions of deaths in what is the deadliest conflict since World War II 1. The last decade has seen the use of rape as a weapon of war in the DRC, where rebels and soldiers subject women, men and children to brutalizing attacks, rape, torture, and mutilation. Survivors of the assault are often further traumatized by infections, disease, poverty, stigma and social isolation.

The US plays a significant role in global health. It is both the largest funder of innovation in global health and the largest donor to care and support programs in sub-Saharan Africa-notably through The US President's Emergency Plan for AIDS Relief (PEPFAR) and responses to humanitarian crisis, such as USAID funded programs in DRC. The effectiveness and sustainability of these efforts are limited by gaps in knowledge of the role of social determinants, such as poverty, social isolation, chronic stress and trauma, and limited access to health care services has on the health of women and families. To begin to address these gaps, our overall goal is to build the science base for large-scale implementation of economic programs to improve the health of survivors of trauma living in man-made and natural disaster settings.

ELIGIBILITY:
Inclusion Criteria:

* household in participating 10 villages with at least one member:

  * 16 years or older,
  * male or female
  * interest in animal husbandry microfinance,
  * vulnerable, including survivor of sexual violence, widow, single mother
  * children under age 18 in the home.

Exclusion Criteria:

* do not live in villages included in study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2011-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline Mental health distress at 18 months | Baseline and 18 months post baseline
  10 villages in rural South Kivu province of DRC will be selected for participation. Sixty-100 households in each village will then be randomized to intervention (receive 1st loan pig) and delayed control (receive offspring from loan pig) groups.
  * Outcome will be measured in both intervention and control villages.
  * Measurement of outcome will use self-report by participating household member.
  * An eligible participant is an adult head of household at least 16 years or older.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Glass, PhD, MPH, RN, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- PAIDEK Microfinance, Bukavu, South Kivu, Republic of the Congo

REFERENCES:
- [Derived] Glass N, Perrin NA, Kohli A, Campbell J, Remy MM. Randomised controlled trial of a livestock productive asset transfer programme to improve economic and health outcomes and reduce intimate partner violence in a postconflict setting. BMJ Glob Health. 2017 Feb 28;2(1):e000165. doi: 10.1136/bmjgh-2016-000165. eCollection 2017. PMID 28589002
- [Derived] Kohli A, Perrin NA, Remy MM, Alfred MB, Arsene KB, Nadine MB, Heri BJ, Clovis MM, Glass N. Adult and adolescent livestock productive asset transfer programmes to improve mental health, economic stability and family and community relationships in rural South Kivu Province, Democratic Republic of Congo: a protocol of a randomised controlled trial. BMJ Open. 2017 Mar 14;7(3):e013612. doi: 10.1136/bmjopen-2016-013612. PMID 28292764
- [Derived] Glass N, Perrin NA, Kohli A, Remy MM. Livestock/animal assets buffer the impact of conflict-related traumatic events on mental health symptoms for rural women. PLoS One. 2014 Nov 24;9(11):e111708. doi: 10.1371/journal.pone.0111708. eCollection 2014. PMID 25419743